CLINICAL TRIAL: NCT01641640
Title: A Phase 3, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of GS-7977 With Peginterferon Alfa 2a and Ribavirin for 12 Weeks in Treatment-Naive Subjects With Chronic Genotype 1, 4, 5, or 6 HCV Infection
Brief Title: Sofosbuvir With Peginterferon Alfa 2a and Ribavirin for 12 Weeks in Treatment-Naive Subjects With Chronic Genotype 1, 4, 5, or 6 HCV Infection
Acronym: NEUTRINO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0110
Record Dates: First submitted 2012-07-09; First posted 2012-07-17 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Hepatitis C
Keywords: HCV genotype 1 (GT-1); HCV genotype 4 (GT-4); HCV genotype 5 (GT-5); HCV genotype 6 (GT-6); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Treatment-Naïve; GS-7977; Ribavirin; RBV; Peginterferon Alfa 2a; PEG
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sofosbuvir+PEG+RBV (Experimental)
  Interventions: Drug: Sofosbuvir; Drug: RBV; Drug: PEG

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribasphere®
Drug: PEG — Pegylated interferon alfa-2a (PEG) 180 μg administered once weekly by subcutaneous injection
  Other Names: PEGASYS®

SUMMARY:
This study was to assess whether sofosbuvir in combination with ribavirin (RBV) and pegylated interferon alfa 2a (PEG) administered for 12 weeks is safe and effective in patients with hepatitis C virus (HCV) genotypes 1, 4, 5 , or 6 as assessed by the rate of sustained viral response (SVR) 12 weeks after discontinuation of therapy (SVR12).

ELIGIBILITY:
Inclusion Criteria:

* Infection with HCV genotype 1, 4, 5, or 6
* Cirrhosis determination
* Subject met the following classifications:

  * Treatment-naive
  * Screening laboratory values within defined thresholds
  * Not treated with any investigational drug or device within 30 days of screening
* Use of highly effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Prior exposure to an direct-acting antiviral targeting the HCV nonstructural protein (NS)5B polymerase
* Pregnant or nursing female, or male with pregnant female partner
* Current or prior history of clinical hepatic decompensation
* History of clinically-significant illness or any other major medical disorder that may have interfered with subject treatment, assessment, or compliance with the protocol
* Excessive alcohol ingestion or significant drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- United States (55):
  - University of Alabama Birmingham, Birmingham, Alabama
  - SCTI Research Foundation, Coronado, California
  - Kaiser Permanente, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Anthony Mills MD, Inc., Los Angeles, California
  - University of California San Diego, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Kaiser Permanente, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Borland-Groover Clinic Baptist, Jacksonville, Florida
  - University of Miami Center for Liver Diseases, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Orlando Immunology Center (ACH), Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - South Florida Center of Gastroenterology, P.A., Wellington, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Infectious Disease Specialist of Atlanta, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Minnesota Gastroenterology, P.A., Saint Paul, Minnesota
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - ID Care, Hillsborough, New Jersey
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Binghamton Gastroenterology Associates, Binghamton, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Inc, Nashville, Tennessee
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Research Specialists of Texas, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Inova Fairfax Hospital Center for Liver Diseases, Falls Church, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc., Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Fundacion De Investigacion De Diego, San Juan, PR, Puerto Rico

REFERENCES:
- [Result] Lawitz E, Mangia A, Wyles D, Rodriguez-Torres M, Hassanein T, Gordon SC, Schultz M, Davis MN, Kayali Z, Reddy KR, Jacobson IM, Kowdley KV, Nyberg L, Subramanian GM, Hyland RH, Arterburn S, Jiang D, McNally J, Brainard D, Symonds WT, McHutchison JG, Sheikh AM, Younossi Z, Gane EJ. Sofosbuvir for previously untreated chronic hepatitis C infection. N Engl J Med. 2013 May 16;368(20):1878-87. doi: 10.1056/NEJMoa1214853. Epub 2013 Apr 23. PMID 23607594
- [Result] Younossi ZM, Stepanova M, Henry L, Gane E, Jacobson IM, Lawitz E, Nelson D, Gerber L, Nader F, Hunt S. Effects of sofosbuvir-based treatment, with and without interferon, on outcome and productivity of patients with chronic hepatitis C. Clin Gastroenterol Hepatol. 2014 Aug;12(8):1349-59.e13. doi: 10.1016/j.cgh.2013.11.032. Epub 2013 Dec 6. PMID 24316172
- [Derived] Stepanova M, Nader F, Cure S, Bourhis F, Hunt S, Younossi ZM. Patients' preferences and health utility assessment with SF-6D and EQ-5D in patients with chronic hepatitis C treated with sofosbuvir regimens. Aliment Pharmacol Ther. 2014 Sep;40(6):676-85. doi: 10.1111/apt.12880. Epub 2014 Jul 15. PMID 25040192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 55 study sites in the United States. The first participant was screened on 18 June 2012. The last participant observation was on 16 April 2013.
Pre-assignment Details: 456 participants were screened and 328 were enrolled; 327 participants were treated, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- Sofosbuvir+PEG+RBV: Participants received Sofosbuvir+pegylated interferon alfa 2a (PEG)+ribavirin (RBV) for 12 weeks and were followed for 24 weeks following treatment.
  Sofosbuvir (400 mg) was administered as an oral tablet, PEG (180 µg) as a subcutaneous injection, and RBV (1000-1200 mg) as 200 mg oral tablets.
Period: Overall Study
Arm/Group | Sofosbuvir+PEG+RBV
Started | 328
Enrolled and Treated | 327
Completed | 292
Not Completed | 36
Not completed — Enrolled but not treated | 1
Not completed — Efficacy failure | 29
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Sofosbuvir+PEG+RBV: Participants received Sofosbuvir+PEG+RBV for 12 weeks and were followed for 24 weeks following treatment.
  Sofosbuvir (400 mg) was administered as an oral tablet, PEG (180 µg) as a subcutaneous injection, and RBV (1000-1200 mg) as 200 mg oral tablets.
Arm/Group | Sofosbuvir+PEG+RBV
Number analyzed (Participants) | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46
  Not Hispanic or Latino | 281
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 54
  White | 257
  Asian | 7
  American Indian/ Alaska Native/ First Nations | 6
  Hawaiian or Pacific Islander | 2
  Other | 1
Hepatitis C Virus (HCV) genotype [Number; unit: participants]
  Genotype 1a/1b | 1
  Genotype 1a | 225
  Genotype 1b | 66
  Genotype 4 | 28
  Genotype 5 | 1
  Genotype 6 | 6
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.4 (0.67)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 71
  ≥ 6 log10 IU/mL | 256
IL28 Genotype [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 95
    CT | 181
    TT | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response (SVR)12
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) 12 weeks after cessation of therapy.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+PEG+RBV
Number analyzed (Participants) | 327
percentage of participants | 91
Statistical Analysis 1: Comparison: Sofosbuvir+PEG+RBV; Superiority would be demonstrated if the SVR12 rate was higher than the 60% null SVR rate based on historical control data; Test type: Superiority or Other; p < 0.001, Binomial exact test

2. Primary Outcome: Number of Participants Experiencing Adverse Events Leading to Permanent Discontinuation of Study Drug
Description: The number of participants experiencing adverse events leading to permanent discontinuation of study drug was summarized. Adverse events may or may not have been related to study treatment. Participants discontinuing study drug were permitted to remain on the study for further assessments.
Time Frame: Baseline to Week 12
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Sofosbuvir+PEG+RBV
Number analyzed (Participants) | 327
participants
  Anaemia | 2
  Haemolytic anaemia | 1
  Neutropenia | 1
  Vision blurred | 1
  Blood creatinine increased | 1
  Haemoglobin abnormal | 1
  Dermatitis | 1

3. Secondary Outcome: Percentage of Participants Achieving SVR4
Description: SVR4 was defined as HCV RNA < LLOQ 4 weeks after cessation of therapy
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+PEG+RBV
Number analyzed (Participants) | 327
percentage of participants | 92.4

4. Secondary Outcome: Percentage of Participants Achieving SVR24
Description: SVR24 was defined as HCV RNA < LLOQ 24 weeks after cessation of therapy
Time Frame: Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+PEG+RBV
Number analyzed (Participants) | 327
percentage of participants | 90.5

5. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment, confirmed with 2 consecutive values (second confirmation value could be posttreatment), or last available on-treatment measurement with no subsequent follow-up values.
Time Frame: Baseline to Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+PEG+RBV
Number analyzed (Participants) | 327
percentage of participants | 0.0

6. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement.
Time Frame: End of treatment to post-treatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir+PEG+RBV
Number analyzed (Participants) | 326
percentage of participants | 8.6

ADVERSE EVENTS:
Time Frame: Baseline to Week 12 plus 30 days
Arm/Group | Sofosbuvir+PEG+RBV
Serious Adverse Events (participants affected / at risk) | 4/327
Other Adverse Events (participants affected / at risk) | 310/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir+PEG+RBV (N=327)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cryoglobulonaemia (Immune system disorders) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir+PEG+RBV (N=327)
Anaemia (Blood and lymphatic system disorders) | 68
Neutropenia (Blood and lymphatic system disorders) | 54
Nausea (Gastrointestinal disorders) | 112
Diarrhoea (Gastrointestinal disorders) | 39
Vomiting (Gastrointestinal disorders) | 39
Constipation (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 194
Pyrexia (General disorders) | 57
Chills (General disorders) | 54
Influenza like illness (General disorders) | 51
Irritability (General disorders) | 43
Pain (General disorders) | 33
Injection site reaction (General disorders) | 27
Injection site erythema (General disorders) | 21
Decreased appetite (Metabolism and nutrition disorders) | 58
Arthralgia (Musculoskeletal and connective tissue disorders) | 47
Myalgia (Musculoskeletal and connective tissue disorders) | 45
Back pain (Musculoskeletal and connective tissue disorders) | 19
Headache (Nervous system disorders) | 118
Dizziness (Nervous system disorders) | 41
Insomnia (Psychiatric disorders) | 81
Depression (Psychiatric disorders) | 31
Anxiety (Psychiatric disorders) | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 34
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 60
Pruritus (Skin and subcutaneous tissue disorders) | 56
Alopecia (Skin and subcutaneous tissue disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years